CLINICAL TRIAL: NCT06137222
Title: Prospective, Multicenter, Randomized, Controlled Clinical Trial of the Tenex Ultrasound System (TXB MicroTip) for Wound Care in Patients With Wagner Type 1-2 Diabetic Foot Ulcers (DFUs)
Brief Title: Prospective, Multicenter, RCT of the Tenex Ultrasound System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tenex Health Inc. (Industry)
Collaborators: Trice Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TenexInc
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU, healing, Wagner Classification
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized controlled clinical trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SOC plus TXB MicroTip Ultrasound (Experimental): Sharp debridement of the outer margins of the index DFU using standard technique (curettage or sharp blade debridement) plus a single additional percutaneous debridement of bone and surrounding tissue via the TXB MicroTip for the first treatment session only plus wound care offloading. The index foot ulcer will be dressed with collagen alginate, gauze and roll gauze. Each subject will return for weekly wound assessment, serial sharp debridement if needed and repeat dressing changes. This care will occur for a duration of 12 weeks or until wound closure is confirmed.
  Interventions: Device: Tenex TXB MicroTip Ultrasound system plus SOC
- SOC (Placebo Comparator): Subcutaneous sharp debridement of the index DFU using standard technique (curettage or sharp blade debridement) plus wound care offloading. The index foot ulcer will be dressed with collagen alginate, gauze and roll gauze. Each subject will return for weekly wound assessment, serial sharp debridement if needed and repeat dressing changes. This care will occur for a duration of 12 weeks or until wound closure is confirmed. Defined as standard of care (SOC).
  Interventions: Other: Standard of Care for diabetic foot ulcer

INTERVENTIONS:
Device: Tenex TXB MicroTip Ultrasound system plus SOC — Subcutaneous sharp debridement of the index DFU using standard technique (curettage or sharp blade debridement) plus wound care offloading. The index foot ulcer will be dressed with collagen alginate, gauze and roll gauze. Each subject will return for weekly wound assessment, serial sharp debridement if needed and repeat dressing changes. This care will occur for a duration of 12 weeks or until wound closure is confirmed. Defined as standard of care (SOC).
  Arms: SOC plus TXB MicroTip Ultrasound
Other: Standard of Care for diabetic foot ulcer — Use of standard of care for the treatment of a diabetic foot ulcer
  Arms: SOC

SUMMARY:
The goal of this multicenter randomized controlled trial is compare standard of care (SOC) to Tenex MicroTip ultrasound therapy plus SOC in patients with Wagner 1-2 diabetic foot ulcers. The main outcomes to answer are:

Does the use of the TXB MicroTip plus SOC increase complete wound healing in Wagner 1-2 diabetic foot ulcer (DFUs) vs. SOC only at 12 weeks (end of treatment)?

Does the use of the TXB MicroTip plus SOC increase complete wound healing in Wagner 1-2 DFUs vs. SOC over a subsequent to treatment 12 month follow-up?

Participants will be asked to come in weekly over a 12 week period for treatment of the Wagner 1-2 DFUs til the DFU is healed. Those whose DFU has healed over the 12 week period will be assessed for durability of healing over a subsequent 12 month period (with assessments occurring monthly.

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to receive either:

• Sharp debridement of the outer margins of the index DFU using standard technique (curettage or sharp blade debridement) plus a single additional percutaneous debridement of bone and surrounding tissue via the TXB MicroTip plus wound care offloading. The index foot ulcer will be dressed with collagen alginate, gauze and roll gauze. Each subject will return for weekly wound assessment, serial sharp debridement if needed and repeat dressing changes. This care will occur for a duration of 12 weeks or until wound closure is confirmed.

OR;

• Subcutaneous sharp debridement of the index DFU using standard technique (curettage or sharp blade debridement) plus wound care offloading. The index foot ulcer will be dressed with collagen alginate, gauze and roll gauze. Each subject will return for weekly wound assessment, serial sharp debridement if needed and repeat dressing changes. This care will occur for a duration of 12 weeks or until wound closure is confirmed. Defined as standard of care (SOC).

Target Population: Adult patients (≥18 years of age) with a documented history of Type 1 or 2 diabetes mellitus (DM) requiring oral and/or insulin replacement therapy and; presenting with Wagner 1- 2 DFUs that are 1 cm2 - 10 cm2 in size.

Duration: The study duration for the individual subject will be at one year follow-up for the determination of recurrence of index site ulceration (upon healing that occurred as part of the 12 weeks of treatment) or; if DFU is not healed at 12 weeks; at the end of 12 weeks of treatment. Note: SOC patients who have not healed at 12 weeks will be offered Tenex therapy over a subsequent 12 week treatment period (i.e. SOC crossed over to Tenex) . If the index ulcer in the crossed over arm heals by 12 weeks, then these healed ulcers will also be followed monthly for a period of 1 year. If the index ulcer in the crossed over patients does not heal in 12 weeks, then they will be defined as such (not healed) and terminated from the trial. All non-healed ulcers will continue to receive treatment as per SOC.

Study Visit Schedule and assessments: Consented subjects at screening will be scheduled for a baseline/treatment initiation visit. The screening visit is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study and consists of a series of screening assessments designed to determine eligibility. Written informed consent is to be obtained prior to obtaining any protected health information and prior to the performance of any protocol specific procedure. Subjects are eligible to enter the Treatment Phase immediately once all the inclusion and none of the exclusion criteria are met. The Investigator will select the study index ulcer of those deemed eligible to proceed. Each subject will have only one DFU selected as the index ulcer. If the subject has more than one DFU at the screening visit, the Investigator will select the largest DFU that meets the eligibility criteria of the protocol as the index ulcer. Eligible consenting subjects will be randomized to either the MicroTip or control group.

Follow-up clinical visits of all enrolled subjects will occur weekly over a 12 week period until either 12 weeks has transpired or; healing of the index ulcer has occurred. Patients will be assessed monthly over 12 months for durability of wound healing of the index ulcer. The 12 month timeframe for follow up will occur at the start of the confirmation of a healed wound.

Investigational Medical Device: The TXB MicroTip imparts low frequency ultrasonic energy by way of the hollow TXB MicroTip that is activated by a foot peddle, irrigates, and cools the TXB MicroTip though an outer sheath and aspirates the debris through the lumen of the hollow TXB MicroTip removing it from the field of treatment. The beveled end of the tip cuts by direct tissue contact. Ultrasonic energy drives the needle and propagates an energy wave in the tissue. Cavitation facilitates rapid pressure changes from ultrasonic vibrations cause small bubbles to form and collapse.

Primary Endpoint: Incidence of index ulcers closed by 12 weeks, where healing has been confirmed 2 weeks after the investigator considers the ulcer healed. The definition of a completely healed DFU is: Intact skin, meaning complete epithelialization without any drainage of a previously ulcerated site .

Primary Safety Endpoint: Incidence of adverse events (AEs) and serious adverse events (SAEs). Adverse events are defined as: mild (asymptomatic or mild symptoms, clinical or diagnostic observation only; intervention not indicated); moderate (local or non-invasive intervention indicated; limitations to age appropriate activities of daily living); serious/severe: death, life threatening, hospitalization or prolongation of hospitalization is indicated, persistent or significantly disabling event. The safety endpoint will be evaluated over a period of 12 weeks of intervention (except for re-ulceration and infection which would be followed for 12 months as defined per below under secondary endpoints).

Medical device deficiencies (of TXB MicroTip) that result in an adverse event (including the causality of intervention as assessed by the clinical judgement of the investigator) or not; are also to be recorded. Device deficiencies include: malfunctions, use errors, and inadequacy of the information provided by the manufacturer.

Re-ulceration of a healed wound during the follow up (12 month phase), will be documented as an adverse event and defined as mild, moderate, or serious/severe as per above.

Secondary Endpoints:

* Percent area reduction of index DFU at 4, 8 and 12 weeks as measured by CarePics (also see Appendix for explanation of CarePics).
* Durability of healing as measured by incidence of re-ulceration within a 12 month follow up period. Note the start of the 12 month timeframe will start upon wound healing at any point during the 12 weeks of treatment.
* Time to healing of those SOC patients who have not healed at 12 weeks if crossed-over to Tenex. Time to healing would be defined when crossed-over (start) and over a subsequent 12 week treatment period. These patients would be followed monthly for 12 months post healing for durability of healing. Healing would be defined as per the primary endpoint above. This cohort of patients will be evaluated as part of the durability of healing endpoint for the Tenex arm as per above and; also separately.
* Incidence of new onset infection of index ulcer (also defined as an adverse event). Infection is to be diagnosed by 2 signs of inflammation or purulence and culture. Infection is also to be graded using the International Working Group Diabetic Foot Ulcer working group (IWGDF) classification system.

ELIGIBILITY:
Key Inclusion Criteria:

1. At least 18 years of age
2. Documented history of Type I or Type II Diabetes Mellitus requiring oral and/or insulin replacement therapy
3. Presence of a DFU Wagner 1 - 2 grade wound on any aspect of the foot, provided it is at or below the medial malleolus.
4. If other wounds are present on the same foot, they must be more than 2 cm distant from the index ulcer.
5. Index ulcer (post-debridement) is a minimum of 1.0 cm2 and a maximum of 10 cm2 at screening visit and treatment visit. The area of the DFU index ulcer is to be measured via the CarePics platform (also see Appendix for explanation of what CarePics does).
6. Adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) measurement of ≥ 30 or an Ankle Branchial Index (ABI) of ≥ 0.7 and ≤ 1.2 or; Arterial Doppler with a minimum of biphasic flow or; Toe Brachial Index (TBI) ≥ 0.75 , using the affected study extremity within 30 days of screening or; great toe pressure >50mmHg.
7. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
8. Properly obtained written informed consent
9. Subject must have stable living environment in order to manage offloading and wound care management.

Key Exclusion Criteria:

1. Index ulcer and/or index limb with presence of gangrene or unstable ischemia at screening and baseline/treatment initiation visit. Note: Baseline/treatment initiation visit should be no more than 10 days after screening. If baseline/treatment initiation visit >10 days after screen, rescreen patient.
2. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids > 10mg prednisone (or equivalent daily dose), cytotoxic chemotherapy, or who are anticipated to require such medications during the study.
3. Index ulcer treated within the last 30 days prior to screening with a prohibited treatment or throughout the trial:

   * Negative pressure therapies
   * Hyperbaric Oxygen
   * Any cellular and/or tissue-based products or wound dressings that include growth factors (e.g., EpiFix®, Regranex, Dermagraft®, Apligraf®, GraftJacket™, OASIS®, PriMatrix®)
4. Active Charcot's arthropathy of the index ulcer limb as verified by clinical evaluation, and/or imaging (x-ray or MRI) within 30 days prior to screening.
5. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence to medical treatment including offloading.
6. Subjects with osteomyelitis on the same limb as the index ulcer as verified by clinical evaluation, and/or imaging (x-ray or MRI) within 30 days prior to screening. Note that with Wagner 1 DFUs, an Xray or MRI would be required for diagnosis of osteomyelitis. For Wagner 2 DFUs, an MRI would be required for diagnosis of osteomyelitis.
7. Presence of diabetes with poor metabolic control as documented with an HbA1c ≥12.0 within 60 days of screening.
8. Subjects with end stage renal disease on hemodialysis.
9. Infected index ulcer at screening. Note: Patient can be rescreened once the infection is deemed clinically resolved.
10. Any clinically significant finding, in the judgment of the investigator, that would place the subject at health risk, impact the study, or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-12-04 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
Wager 1-2 DFU healing. Primary outcome endpoint. | 12 weeks
  Incidence of index ulcers closed by 12 weeks, where healing has been confirmed 2 weeks after the investigator considers the ulcer healed. The definition of a completely healed DFU is: Intact skin, meaning complete epithelialization without any drainage of a previously ulcerated site
Incidence of adverse events (AEs) and serious adverse events (SAEs). Primary safety endpoint | 12 weeks
  Adverse events are defined as: mild (asymptomatic or mild symptoms, clinical or diagnostic observation only; intervention not indicated); moderate (local or non-invasive intervention indicated; limitations to age appropriate activities of daily living); serious/severe: death, life threatening, hospitalization or prolongation of hospitalization is indicated, persistent or significantly disabling event

SECONDARY OUTCOMES:
Durability of healing as measured by incidence of re-ulceration within a 12 month follow up period. | 12 months
  Number of completely healed wounds @ 12 weeks that re-ulcerate over a 12 month period.
Wound size (area in cm2) reduction from baseline/treatment initiation | 12 weeks
  Evaluate:
  * Wound area reduction from baseline/treatment initiation at 4 weeks
  * Wound area reduction from baseline/treatment initiation at 8 weeks.
  * Wound area reduction from baseline/treatment initiation at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Van Gils, DPM, Principal Investigator — St. George Regional Hospital
Locations (2):
- United States (2):
  - Springhill Medical Center, Mobile, Alabama
  - St. George Regional Hospital, St. George, Utah

IPD SHARING:
Plan to Share IPD: Undecided